CLINICAL TRIAL: NCT02341534
Title: BIO monitorinG in Patients With Preserved Left ventricUlar Function AfteR Diagnosed Myocardial Infarction
Acronym: BIO-GUARD-MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Collaborators: IHF GmbH - Institut für Herzinfarktforschung (Other); Qmed Consulting A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HS058; Preserved Ejection Fraction (Other: BIOTRONIK); Implantable Cardiac Device (Other: BIOTRONIK); Loop Recorder (Other: BIOTRONIK); ICM (Other: BIOTRONIK)
Record Dates: First submitted 2014-12-12; First posted 2015-01-19 (Estimated); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Infarction; Myocardial Infarction, Acute; Myocardial Infarction Old
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent Endpoint Committee was installed to evaluate all reported cardiovascular and serious AEs. The information provided to the Committee did not contain information about the group assigment of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BioMonitor arm (Other): BioMonitor group (implantation with investigational device + transfer of information via Home Monitoring)
  Interventions: Device: BioMonitor
- Control arm (No Intervention): Control group (standard of care)

INTERVENTIONS:
Device: BioMonitor — Patients will be implanted with the BioMonitor + Home Monitoring feature
  Arms: BioMonitor arm

SUMMARY:
The BIO|GUARD-MI study investigates whether continuous arrhythmia monitoring and the consequent treatment after detected arrhythmias in patients after myocardial infarction with preserved cardiac function, but other risk factors, decreases the risk of major adverse cardiac events.

DETAILED DESCRIPTION:
Patients randomized to the BioMonitor arm will receive an implantable cardiac monitor (ICM; BioMonitor) with remote monitoring function (Home Monitoring®). If the device detects and reports an arrhythmia, patients will be appropriately examined and treated. Patients randomized to the control arm will receive best proven treatment, but no implantable cardiac monitor.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of MI according to guidelines
* CHA2DS2-VASc-Score ≥ 4 in men / ≥ 5 in women
* LVEF > 35 % as estimated within 6 months before enrollment but after conclusion of AMI treatment
* Patient accepts activation of Home Monitoring®
* Patient is able to understand the nature of the clinical study and has provided written informed consent

Exclusion Criteria:

* Patients with hemorrhagic diathesis
* Permanent oral anticoagulation treatment for atrial fibrillation
* Indication for chronic renal dialysis
* Pacemaker or ICD implanted or indication for implantation
* Parkinson's disease
* Life expectancy < 1 year
* Participation in another interventional clinical Investigation
* Age < 18 years
* Woman who are pregnant or breast feeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jons, Doctor, Study Chair — Rigshospitalet; Denmark; Copenhagen; Steffen Behrens, Professor, Principal Investigator — Vivantes Humboldt Klinikum, Germany, Berlin; Poul Erik Bloch Thomsen, Professor, Study Director — Aalborg University Hospital, Denmark, Aalborg; Peter Sogaard, Professor, Principal Investigator — Aalborg University Hospital, Denmark, Aalborg
Locations (59):
- United States (8):
  - Gateway Cardiology, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Altru Health System, Grand Forks, North Dakota
  - Abington Medical Specialists, Abington, Pennsylvania
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Carolina Cardiology Associates, Rock Hill, South Carolina
  - Metro Knoxville HMA LLC, Knoxville, Tennessee
- Australia (3):
  - Lyell McEwin Hospital (LMH), Elizabeth Vale, South Australia
  - East Metropolitan Health Service Trading AS Royal Perth HOSPITAL, Perth, Western Australia
  - The Canberra Hospital, Canberra
- Kepler Universitätsklinikum, Linz, Upper Austria, Austria
- Belgium (2):
  - OLV Ziekenhuis Aalst, Aalst
  - Ziekenhuis Oost Limburg Genk (ZOL Genk), Genk
- Czechia (3):
  - Nemocnice České Budějovice, České Budějovice
  - Fakultní nemocnice Olomouc, Olomouc
  - Institute for Clinical and Experimental Medicine (IKEM), Prague
- Denmark (7):
  - Odense University Hospital (OUH), Odense, Region Syddanmark
  - Aalborg Universitetshospitel, Aalborg
  - Århus Universitetshospital, Århus N
  - Rigshospitalet, Copenhagen
  - Regionshospitalet Herning, Herning
  - Sjaellands Universitets Hospital, Roskilde, Roskilde
  - Regionshospitalet Viborg, Viborg
- France (2):
  - CHRU de Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Hôpital Gabriel Montpied, Clermont Ferrand, Clermont-Ferrand
- Germany (16):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz- und Gefäß- Klinik GmbH Bad Neustadt, Bad Neustadt A.d. Saale
  - Charité Universitätsklinikum - Campus Benjamin Franklin, Berlin
  - Vivantes Humboldt-Klinikum, Berlin
  - Vivantes-Krankenhaus Spandau, Berlin
  - Städtisches Krankenhaus Bielefeld-Mitte, Bielefeld
  - Klinikum Coburg, Coburg
  - Klinikum Fürth, Fürth
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Klinikum der Universität Jena, Jena
  - Herzzentrum Leipzig GmbH, Leipzig
  - Universitätsklinikum Schleswig-Holstein (UKSH) - Campus Lübeck, Lübeck
  - Johannes Wesling Klinikum Minden, Minden
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (6):
  - National Hospital of Cardiology, Balatonfüred
  - Gottsegen György, Budapest
  - Semmelweis Medical University, Budapest
  - Hungarian Defence Forces Military Hospital, Budapest
  - The Debrecen University of Medicine, Debrecen
  - The University of Pécs, Pécs
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis Amsterdam (OLVG), Amsterdam
  - Scheperziekenhuis, Treant Zorggroep, Emmen
- Poland (2):
  - Klinika i Katedra Chorób Wewn. i Kardiologii, Warsaw
  - National Institute of Cardiology, Warsaw
- Slovakia (2):
  - SÚSCCH, Banská Bystrica
  - East-Slovak Cardiology Institute (VUSCH), Košice
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital de la Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

REFERENCES:
- [Derived] Jons C, Bloch Thomsen PE, Riahi S, Smilde T, Bach U, Jacobsen PK, Taborsky M, Falukozy J, Wiemer M, Christensen PD, Konyi A, Schelfaut D, Bulava A, Grabowski M, Merkely B, Nuyens D, Mahajan R, Nagel P, Tilz R, Malczynski J, Steinwender C, Brachmann J, Serota H, Schrader J, Behrens S, Sogaard P. Arrhythmia monitoring and outcome after myocardial infarction (BIO|GUARD-MI): a randomized trial. Front Cardiovasc Med. 2024 May 13;11:1300074. doi: 10.3389/fcvm.2024.1300074. eCollection 2024. PMID 38807948
- [Derived] Jons C, Sogaard P, Behrens S, Schrader J, Mrosk S, Bloch Thomsen PE. The clinical effect of arrhythmia monitoring after myocardial infarction (BIO-GUARD|MI):study protocol for a randomized controlled trial. Trials. 2019 Sep 11;20(1):563. doi: 10.1186/s13063-019-3644-5. PMID 31511057

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 802 patients were enrolled, 12 exited the study before randomization.
Groups:
- BioMonitor Arm: Patients are implanted with investigational device. Device transfers daily arrhythmia information. Investigators react on information if required. If no arrhythmias are detected, patients are followed by standard post-MI routine.
- Control Arm: Patients do not receive investigational device, i.e. no additional arrhythmia monitoring. Patients are followed by standard post-MI routine.
Period: Overall Study
Arm/Group | BioMonitor Arm | Control Arm
Started | 398 | 392
Completed | 322 | 325
Not Completed | 76 | 67

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BioMonitor Arm | Control Arm | Total
Number analyzed (Participants) | 398 | 392 | 790
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (7.7) | 70.8 (8.5) | 71.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 115 | 222
  Male | 291 | 277 | 568
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Major Adverse Cardiac Event (MACE)
Description: The primary endpoint is defined as death for cardiovascular reasons or unplanned hospitalization for cardiovascular reasons as per study protocol.
  The time period with regards to the Time-to-Event Outcome Measures starts with the randomization of the patient.
  All patients will be assessed for Time-to-Event Outcome Measures until formal study termination is announced or until the individual patient meets a drop out criterion in accordance with the study protocol. The study period is estimated 6 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 21.6 [17.7 to 26.2] | 24.3 [20.3 to 29.0]
Statistical Analysis 1: Comparison: BioMonitor Arm vs Control Arm; Test type: Superiority; p = 0.21, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.10]

2. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Outcome of Death Due to Any Cause
Description: The occurrence of death due to any cause will be recorded and analyzed.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 6.7 [4.6 to 9.8] | 7.1 [4.9 to 10.3]

3. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Outcome of Death Due to Any Cause or Heart Transplantation
Description: Assessment of the time from randomization to death for any reason or heart transplantation during the clinical investigation.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 6.7 [4.6 to 9.8] | 7.1 [4.9 to 10.3]

4. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Outcome of Cardiovascular Death or Heart Transplantation
Description: Assessment of the time from randomization to cardiovascular death or heart transplantation during the clinical investigation. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 3.5 [2.1 to 6.0] | 4.7 [2.9 to 7.4]

5. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Worsening of Heart Failure Requiring Hospitalization or Urgent Visit
Description: Assessment of the time from randomization to first hospitalization or urgent visit for worsening of the patient status due to heart failure, or death due to heart failure. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 6.0 [4.0 to 9.0] | 5.9 [3.9 to 8.9]

6. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With an Arrhythmia Resulting in Hospitalization
Description: Assessment of the time from randomization to the first hospitalization resulting from an arrhythmia or death resulting from arrhythmia. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 3.3 [1.8 to 5.9] | 3.4 [2.0 to 5.9]

7. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Acute Coronary Syndrome Resulting in Hospitalization
Description: Assessment of the time from randomization to the first hospitalization resulting from acute coronary syndrome or death resulting from acute coronary syndrome. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 10.6 [7.8 to 14.3] | 15.1 [11.8 to 19.2]

8. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Stroke Resulting in Hospitalization
Description: Assessment of the time from randomization to the first hospitalization resulting from stroke or death resulting from stroke. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 3.6 [2.1 to 6.1] | 3.0 [1.6 to 5.3]

9. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Major Bleeding Resulting in Hospitalization
Description: Assessment of the time from randomization to the first hospitalization resulting from major bleeding or death resulting from major bleeding. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 0.6 [0.2 to 2.4] | 1.1 [0.4 to 2.9]

10. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With Systemic Embolism Resulting in Hospitalization
Description: Assessment of the time from randomization to the first hospitalization resulting from systemic embolism or death resulting from systemic embolism. A specified endpoint definition will be given by the members of the EAEC and documented in the charter agreement.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 0.3 [0 to 2.0] | 0.7 [0.2 to 2.7]

11. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants With an Arrhythmia
Description: Assessment of the time from randomization to first arrhythmia.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 53.6 [48.5 to 58.8] | 10 [7.3 to 13.5]

12. Secondary Outcome: Type of Initiated Therapies
Description: Post-hoc categorical summary of most frequent therapies initiated after detection of arrhythmias.
Time Frame: All data are collected for the period from randomization until official study end or drop-out, for all enrolled patients, up to 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 195 | 44
Participants
  Oral anticoagulation treatment | 84 | 18
  Pacemaker implantation | 45 | 6
  Reduction of heart-rate lowering drugs | 43 | 5
  Betablocker treatment | 13 | 6
  Antiarrhythmics | 10 | 9

13. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants Receiving Therapy After Arrhythmia Diagnosis
Description: Assessment of the time from randomization to first therapy. In this context therapy is the attempted remediation of the patient's regular heartbeat.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
percentage of patients with event | 53.6 [48.5 to 58.8] | 10.0 [7.3 to 13.5]

14. Secondary Outcome: Change in World Health Organization Five Well-being Index (WHO-5) From 6 Months to 24 Months.
Description: A further secondary endpoint is the assessment of the patient's well-being. The patient's well-being will be recorded during the regular telephone contacts using the WHO-5 Well-being Index. The scale reaches from 0 (worst status) to 100 (best possible status).
Time Frame: We report the intraindividual change from 6-months to 24-months. All data are collected for the period from randomization until official study end or drop-out, for all enrolled patients.
Measure: Mean (Standard Deviation); unit: Change in units on the WHO-5 scale
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 398 | 392
Change in units on the WHO-5 scale | 0.1 (17.6) | 0.7 (21.2)

15. Other Pre Specified Outcome: Mean Value of EQ-5D-5L
Description: The EQ-5D-5L questionnaire was administered during the telephone contacts to estimate utility values at different time points for an economic evaluation.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The scale reaches from 0 (worst status) to 100 (best possible status).
Time Frame: From Baseline measurement to 60 months. All data are collected for the period from randomization until official study end or drop-out, for all enrolled patients.
Population: Not all patients contributed to this endpoint. The EQ-5D-5L was only introduced later in the trial via an amendment in 2019.
Measure: Mean (Standard Deviation); unit: Units on the EQ-5D-5L scale
Arm/Group | BioMonitor Arm | Control Arm
Number analyzed (Participants) | 353 | 351
Units on the EQ-5D-5L scale
  Baseline: number analyzed (Participants) | 89 | 81
  Baseline | 74.9 (16.4) | 75.0 (18.8)
  12-months: number analyzed (Participants) | 162 | 151
  12-months | 72.5 (17.7) | 73.2 (16.9)
  24-months: number analyzed (Participants) | 147 | 141
  24-months | 71.6 (18.2) | 71.3 (18.1)
  36-months: number analyzed (Participants) | 110 | 114
  36-months | 71.2 (19.2) | 69.5 (18.4)
  48-months: number analyzed (Participants) | 66 | 71
  48-months | 69.9 (17.3) | 69.8 (19.2)
  60-months: number analyzed (Participants) | 15 | 17
  60-months | 74.8 (20.8) | 64.4 (21.2)

ADVERSE EVENTS:
Time Frame: 2 years and 9 months mean follow-up duration
Description: Adverse event definitions in this trial are based on ISO14155.
Arm/Group | BioMonitor Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 43/398 | 42/392
Serious Adverse Events (participants affected / at risk) | 300/398 | 267/392
Other Adverse Events (participants affected / at risk) | 259/398 | 173/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioMonitor Arm (N=398) | Control Arm (N=392)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 3 (3) | 2 (2)
Abscess rupture (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 10 (12)
Acute myocardial infarction (Cardiac disorders) | 27 (30) | 35 (44)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 24 (30) | 15 (20)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol interaction (General disorders) | 0 (0) | 1 (1)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Ammonia increased (Investigations) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 8 (10)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 18 (20) | 27 (36)
Angina unstable (Cardiac disorders) | 3 (3) | 15 (17)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 1 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 3 (3)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 4 (4)
Aortic valve calcification (Cardiac disorders) | 0 (0) | 3 (3)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 5 (5) | 3 (4)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 4 (4) | 4 (4)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (3) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Atheroembolism (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 65 (71) | 25 (32)
Atrial flutter (Cardiac disorders) | 9 (9) | 6 (6)
Atrial pressure increased (Investigations) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 3 (4)
Atrioventricular block (Cardiac disorders) | 6 (6) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 11 (11) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 9 (10) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (4) | 4 (4)
Benign tracheal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister infected (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood electrolytes decreased (Investigations) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 4 (4) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 3 (3)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bundle branch block left (Cardiac disorders) | 4 (4) | 5 (5)
Bundle branch block right (Cardiac disorders) | 2 (2) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 2 (2)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 12 (12) | 8 (8)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 25 (37) | 32 (52)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac failure high output (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve abscess (Infections and infestations) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 2 (2)
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 3 (3)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 7 (7) | 2 (2)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 6 (6) | 5 (5)
Cataract (Eye disorders) | 8 (10) | 14 (16)
Cataract diabetic (Eye disorders) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis pharyngeal (Infections and infestations) | 1 (1) | 0 (0)
Central auditory processing disorder (Nervous system disorders) | 0 (0) | 1 (1)
Central pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 4 (4) | 3 (3)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 10 (10) | 9 (11)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 2 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (2)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest pain (General disorders) | 11 (11) | 10 (14)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 11 (12)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 8 (8)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chorea (Nervous system disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (25) | 11 (14)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 6 (6)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Community acquired infection (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Condition aggravated (General disorders) | 15 (16) | 15 (17)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (5) | 3 (3)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 2 (3)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Corona virus infection (Infections and infestations) | 11 (11) | 13 (13)
Coronary artery disease (Cardiac disorders) | 11 (11) | 18 (20)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 4 (4)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 19 (24) | 24 (25)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Crepitations (General disorders) | 2 (2) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 2 (2)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cystitis escherichia (Infections and infestations) | 0 (0) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Death (General disorders) | 5 (5) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 11 (14) | 7 (8)
Delirium (Psychiatric disorders) | 4 (4) | 3 (3)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Device battery issue (Product Issues) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 1 (1)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Device pacing issue (Product Issues) | 1 (1) | 0 (0)
Device psychogenic complication (General disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Diabetic blindness (Eye disorders) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1)
Disease recurrence (General disorders) | 0 (0) | 1 (1)
Dislocation of sternum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Disorganised speech (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 3 (3)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 7 (8) | 6 (7)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Duodenal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 10 (15)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Echocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Ectropion (Eye disorders) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 2 (2) | 6 (6)
Electrocardiogram ST segment depression (Investigations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 2 (2) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 5 (5) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Exposure to chemical pollution (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to violent event (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 19 (21) | 20 (21)
Fatigue (General disorders) | 3 (3) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Food refusal (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Gallbladder enlargement (Hepatobiliary disorders) | 0 (0) | 1 (2)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 6 (6)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4)
General physical health deterioration (General disorders) | 9 (9) | 8 (8)
General symptom (General disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 3 (4)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 4 (4)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 2 (2)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (4)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 6 (6) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 15 (16) | 6 (6)
Hypertensive crisis (Vascular disorders) | 8 (16) | 9 (11)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hypotension (Vascular disorders) | 8 (8) | 4 (4)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 2 (2) | 1 (1)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Implant site abscess (Infections and infestations) | 1 (1) | 0 (0)
Implant site dehiscence (General disorders) | 4 (4) | 0 (0)
Implant site erosion (General disorders) | 3 (3) | 0 (0)
Implant site haematoma (General disorders) | 2 (2) | 0 (0)
Implant site haemorrhage (General disorders) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 7 (7) | 0 (0)
Implant site irritation (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 3 (3) | 0 (0)
Implant site swelling (General disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 5 (6) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 6 (6) | 3 (3)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 4 (5) | 5 (6)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Investigation noncompliance (Social circumstances) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 4 (4)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Klebsiella infection (Infections and infestations) | 2 (2) | 1 (1)
Lacunar infarction (Nervous system disorders) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 7 (7) | 2 (2)
Laryngeal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 4 (4) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (4) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 8 (8)
Loss of personal independence in daily activities (Social circumstances) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 4 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphatic fistula (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 2 (2) | 0 (0)
Maisonneuve fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 4 (4)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical device site fistula (General disorders) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to muscle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Mononuclear cell count increased (Investigations) | 1 (1) | 0 (0)
Morganella infection (Infections and infestations) | 0 (0) | 1 (1)
Multimorbidity (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 4 (4)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 6 (7) | 6 (6)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 6 (7)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 3 (5)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
No adverse event (General disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 4 (5)
Normal tension glaucoma (Eye disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Nosocomial infection (Infections and infestations) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 5 (5) | 1 (1)
Oesophageal adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Organ failure (General disorders) | 1 (1) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 2 (2)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (7)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (1)
Pain (General disorders) | 5 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 2 (2) | 0 (0)
Pathogen resistance (Infections and infestations) | 2 (2) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (12) | 11 (14)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 3 (3) | 2 (4)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 4 (5) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (3)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 3 (3)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 15 (16)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 30 (35) | 28 (37)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 4 (4) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (3)
Polyp (General disorders) | 3 (3) | 2 (2)
Porcelain gallbladder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postoperative hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 2 (2)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 4 (4) | 0 (0)
Product administration interrupted (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Protein deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pseudolymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Raoultella test positive (Investigations) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Refusal of treatment by patient (Social circumstances) | 0 (0) | 1 (1)
Renal aneurysm (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal atrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 4 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 4 (4)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 6 (6) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 5 (5)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 4 (5)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Salivary gland calculus (Gastrointestinal disorders) | 1 (2) | 1 (1)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (3)
Sepsis (Infections and infestations) | 6 (8) | 5 (5)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 2 (2) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 4 (4) | 1 (1)
Sinus arrest (Cardiac disorders) | 13 (14) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 10 (10) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 17 (18) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Snapping hip syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0)
Stomatitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 3 (3)
Subclavian artery stenosis (Vascular disorders) | 2 (2) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Sudden death (General disorders) | 0 (0) | 1 (1)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 3 (4)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 11 (12) | 11 (14)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (4)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Terminal state (General disorders) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth pulp haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 6 (7) | 4 (4)
Transitional cell cancer of the renal pelvis and ureter localised (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Treatment noncompliance (General disorders) | 0 (0) | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 3 (3) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 5 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 11 (15) | 13 (19)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 2 (2)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (4)
Vascular access site infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular pain (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular stent stenosis (General disorders) | 6 (8) | 15 (17)
Vascular stent thrombosis (General disorders) | 0 (0) | 2 (2)
Vascular wall hypertrophy (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 4 (6)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 13 (15) | 4 (4)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vocal cord scarring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3)
Weight decreased (Investigations) | 4 (5) | 1 (1)
Weight increased (Investigations) | 3 (3) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioMonitor Arm (N=398) | Control Arm (N=392)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Accident at work (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acquired foramen magnum stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 59 (68) | 32 (38)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anal fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 17 (21) | 18 (19)
Angina unstable (Cardiac disorders) | 4 (4) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Aortic dilatation (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arterial fibrosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 48 (60) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 7 (8) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 8 (10) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Auditory disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 12 (12)
Balance disorder (Nervous system disorders) | 2 (2) | 2 (2)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Bile acid malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder hypertrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 2 (2)
Blood pressure decreased (Investigations) | 1 (1) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 24 (26) | 5 (5)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Bundle branch block (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 2 (2) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 14 (14) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (3)
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 16 (17) | 13 (15)
Chills (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 10 (10) | 5 (5)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 5 (6) | 1 (1)
Corona virus infection (Infections and infestations) | 7 (7) | 3 (3)
Coronary artery disease (Cardiac disorders) | 3 (3) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (8)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 5 (5)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Device battery issue (Product Issues) | 6 (6) | 0 (0)
Device dislocation (Product Issues) | 3 (3) | 0 (0)
Device extrusion (Product Issues) | 2 (2) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Discomfort (General disorders) | 1 (1) | 0 (0)
Dislocation of sternum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 16 (18) | 9 (11)
Dizziness postural (Nervous system disorders) | 2 (2) | 0 (0)
Drug therapeutic incompatibility (General disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysbiosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysgraphia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 13 (14)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Ectopic gastric mucosa (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Excessive exercise (Social circumstances) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 3 (3)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 21 (24) | 9 (10)
Fatigue (General disorders) | 6 (6) | 1 (1)
Feeling abnormal (General disorders) | 2 (2) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric mucosa erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric mucosal hypertrophy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal melanosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 5 (5) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Heart rate increased (Investigations) | 2 (2) | 0 (0)
Heart rate irregular (Investigations) | 4 (4) | 0 (0)
Heart valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hernia (General disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 6 (7)
Hypertensive crisis (Vascular disorders) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 4 (4) | 7 (8)
Hypothyroidism (Endocrine disorders) | 0 (0) | 4 (4)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Hypotonic urinary bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Implant site dehiscence (General disorders) | 1 (1) | 0 (0)
Implant site discharge (General disorders) | 1 (1) | 1 (1)
Implant site erythema (General disorders) | 2 (2) | 0 (0)
Implant site haematoma (General disorders) | 5 (5) | 0 (0)
Implant site haemorrhage (General disorders) | 3 (3) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Implant site inflammation (General disorders) | 1 (1) | 0 (0)
Implant site irritation (General disorders) | 2 (2) | 0 (0)
Implant site pain (General disorders) | 6 (6) | 0 (0)
Implant site pruritus (General disorders) | 1 (1) | 0 (0)
Implant site swelling (General disorders) | 2 (2) | 0 (0)
Implant site vesicles (General disorders) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Infarction (Vascular disorders) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 2 (2) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Left atrial dilatation (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (5) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (2) | 1 (1)
Loss of control of legs (General disorders) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lymph node calcification (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (4) | 2 (2)
Medical device discomfort (General disorders) | 3 (3) | 0 (0)
Medical device site irritation (General disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 2 (2)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle oedema (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal abscess (Infections and infestations) | 1 (1) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
New DPC required (Product Issues) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 3 (3) | 2 (2)
Nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Nodal rhythm (Cardiac disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 8 (9) | 10 (10)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 6 (6) | 7 (7)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 2 (2)
Osteitis condensans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (6)
Palpitations (Cardiac disorders) | 3 (3) | 3 (4)
Pancreatic steatosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (2) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Patient dissatisfaction with device (Social circumstances) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
Peripheral venous disease (Vascular disorders) | 2 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 6 (6) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Puncture site infection (Infections and infestations) | 1 (1) | 0 (0)
Purine metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal artery arteriosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal atrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal disorder (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal impairment (Renal and urinary disorders) | 4 (4) | 0 (0)
Renal ischaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal vessel disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 3 (3) | 0 (0)
Sinus arrest (Cardiac disorders) | 14 (15) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 36 (43) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 9 (9) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 12 (13) | 0 (0)
Syncope (Nervous system disorders) | 4 (5) | 3 (3)
Temporal arteritis (Vascular disorders) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thyroid cyst (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tobacco abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 2 (3)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tympanosclerosis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Undersensing (Product Issues) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urogenital atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vascular skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 11 (11) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 24 (27) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 3 (3) | 2 (2)
Weight increased (Investigations) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Study Protocol used in the USA (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT02341534/Prot_000.pdf
  • Study Protocol: Modification to study protocol used in the USA (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT02341534/Prot_001.pdf
  • Study Protocol: Study Protocol used outside the USA (OUS) (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT02341534/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT02341534/SAP_003.pdf